CLINICAL TRIAL: NCT02492178
Title: Bio-availability of Rectal Artesunate in Children With Severe Falciparum Malaria
Acronym: REACH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Kinshasa School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: REACH
Record Dates: First submitted 2015-06-22; First posted 2015-07-08 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IR artesunate + IV artesunate (Experimental): Patients receive 1 dose of intrarectal artesunate (10 mg/ kg b.w.) on admission and 1 dose of intravenous artesunate (2.4 mg/kg body weight) at 12 hours. All patients receive a loading dose of intravenous quinine (20 mg salt/kg b.w.) on admission followed by 10 mg/kg b.w. at 8 and 16 hrs.
  Interventions: Drug: Intrarectal artesunate; Drug: Intravenous artesunate; Drug: Intravenous quinine
- IV artesunate + IR artesunate (Experimental): Patients receive 1 dose of intravenous artesunate (2.4 mg/kg b.w) on admission and 1 dose of intrarectal artesunate (10 mg/ kg b.w.) at 12 hours. All patients receive a loading dose of intravenous quinine (20 mg salt/kg b.w.) on admission followed by 10 mg/kg b.w. at 8 and 16 hrs.
  Interventions: Drug: Intrarectal artesunate; Drug: Intravenous artesunate; Drug: Intravenous quinine

INTERVENTIONS:
Drug: Intrarectal artesunate
  Other Names: artesunate suppositories
Drug: Intravenous artesunate
  Other Names: parenteral artesunate
Drug: Intravenous quinine
  Other Names: parenteral quinine

SUMMARY:
The study aims at describing the pharmacokinetic properties of rectal artesunate in well characterized severely ill patients using intravenous artesunate as a comparator.

DETAILED DESCRIPTION:
Individually randomized, open label, 2-arm, cross-over, clinical trial. Patients are allocated to receive rectal artesunate at admission and intravenous artesunate after 12 hours or intravenous artesunate at admission and rectal artesunate after 12 hours. All patients are treated for severe malaria with intravenous quinine. Frequent blood samples are taken at fixed intervals after the administration of the first and the second dose of study drug. The time frame is 24 hours and thereafter patients continue the standard antimalarial therapy.

ELIGIBILITY:
Inclusion Criteria:

* Weight ≥6 kilograms and ≤ 34 kilograms
* Severe malaria (WHO Guidelines 2013; Appendix 1)
* P. falciparum infection confirmed by Rapid Diagnostic Test (P. falciparum monoinfection or mixed infection with P. ovale or P. malariae)
* Parents or guardian signed Informed Consent

Exclusion Criteria:

* Acute diarrhoea defined as > 3 liquid stools in the previous 24 hours
* Visible anorectal malformations or a disease of the rectum
* Known hypersensitivity to quinine or artesunate
* A documented history of an effective dose of parenteral antimalarial in the preceding 24 hours or a single dose of rectal artesunate in the previous 12 hours or a dose of an artemisinin based combination therapy in the previous 6 hours
* Co-morbidity which in the judgement of the investigator would interfere with the patient treatment or results of the study or place the subject at undue risk
* Participation in another clinical trial or earlier in the same clinical trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2015-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics profile of rectal artesunate | 24 hours
  The pharmacokinetics profile of rectal artesunate (the study drug), consisting of: area under the concentration-time curve; terminal elimination half-life; elimination clearance; apparent volume of distribution will be measured and compared to the pharmacokinetic profile of intravenous artesunate (the comparator).

CONTACTS AND LOCATIONS:
Locations (1):
- Kinshasa School of Public Health, Kinshasa, Democratic Republic of the Congo

REFERENCES:
- [Derived] Fanello C, Hoglund RM, Lee SJ, Kayembe D, Ndjowo P, Kabedi C, Badjanga BB, Niamyim P, Tarning J, Woodrow C, Gomes M, Day NP, White NJ, Onyamboko MA. Pharmacokinetic Study of Rectal Artesunate in Children with Severe Malaria in Africa. Antimicrob Agents Chemother. 2021 Mar 18;65(4):e02223-20. doi: 10.1128/AAC.02223-20. Print 2021 Mar 18. PMID 33526485